CLINICAL TRIAL: NCT05967481
Title: Investigating the Clinical Trial Journey and Engagement of Neuroendocrine Tumor Patients
Brief Title: Evaluation of Study Experiences of Neuroendocrine Tumor Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84454037
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Neuroendocrine Tumors
Keywords: neuroendocrine tumor
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in clinical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This research will admit a wide range of data on the clinical study experience of neuroendocrine tumor patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future patients with neuroendocrine tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of neuroendocrine tumor
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Enrolled in another research study
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuroendocrine tumor who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in a neuroendocrine tumor clinical research | 3 months
Number of neuroendocrine tumor patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walter T, Krzyzanowska MK. Quality of clinical trials in gastroenteropancreatic neuroendocrine tumours. Neuroendocrinology. 2012;96(3):238-48. doi: 10.1159/000337662. Epub 2012 Aug 28. PMID 22414794
- [Background] Faggiano A, Malandrino P, Modica R, Agrimi D, Aversano M, Bassi V, Giordano EA, Guarnotta V, Logoluso FA, Messina E, Nicastro V, Nuzzo V, Sciaraffia M, Colao A. Efficacy and Safety of Everolimus in Extrapancreatic Neuroendocrine Tumor: A Comprehensive Review of Literature. Oncologist. 2016 Jul;21(7):875-86. doi: 10.1634/theoncologist.2015-0420. Epub 2016 Apr 6. PMID 27053503
- [Background] Capdevila J, Teule A, Barriuso J, Castellano D, Lopez C, Manzano JL, Alonso V, Garcia-Carbonero R, Dotor E, Matos I, Custodio A, Casanovas O, Salazar R; EVERLAR study investigators. Phase II Study of Everolimus and Octreotide LAR in Patients with Nonfunctioning Gastrointestinal Neuroendocrine Tumors: The GETNE1003_EVERLAR Study. Oncologist. 2019 Jan;24(1):38-46. doi: 10.1634/theoncologist.2017-0622. Epub 2018 May 23. PMID 29794066

DOCUMENTS (1):
  • Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05967481/ICF_000.pdf